CLINICAL TRIAL: NCT02304640
Title: Prevalence, Severity and Determinants of Cancer-related Fatigue (CRF) in Asian Breast Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Alexandre Chan, Associate Professor and Specialist Pharmacist (Oncology Pharmacy), National University of Singapore
Other Study IDs: 2014/754/B
Record Dates: First submitted 2014-11-21; First posted 2014-12-02 (Estimated); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Fatigue; Chemotherapy; Breast Cancer; Supportive Care
Keywords: fatigue; chemotherapy; breast cancer; supportive care; Singapore
MeSH Terms: conditions — Fatigue; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Early-stage breast cancer patients
- Healthy control

SUMMARY:
There is a paucity of studies that focus on the symptom burden of cancer patients in Singapore, particularly the clinical effects of cancer-related fatigue (CRF). Knowing that early-stage breast cancer is curable, it is of paramount importance to evaluate the clinical and biological determinants of lingering symptoms in breast cancer survivors so that appropriate psychosocial interventions can be formulated.

DETAILED DESCRIPTION:
The investigators hypothesize that variations in clinical and biological determinants contribute to different severities of CRF among Asian breast cancer patients. Through this study, the investigators aim to evaluate the prevalence and severity of CRF among Asian breast cancer patients, and to identify the biological and clinical determinants of CRF among these patients.

This will be a multicenter, prospective, longitudinal, observational study conducted at the National Cancer Centre Singapore and KK Women's and Children's Hospital. Informed consent will be obtained from participants before the investigators proceed with data collection.

The study participants will be assessed at relevant time points. Biological determinants and symptoms associated with CRF will be assessed. The associations between changes in CRF, plasma cytokines levels, serum cortisol levels, and other clinical determinants will be elucidated.

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years of age
* Stage I-III breast cancer
* Chinese, Malay or Indian ethnics
* Surgical treatment has been performed
* Scheduled to receive four cycles of chemotherapy (doxorubicin/cyclophosphamide [AC], docetaxel/cyclophosphamide [TC], 5-fluorouracil/epirubicin/cyclophosphamide [FEC]) (total duration of 3 months) and/or radiotherapy and/or hormonal therapy
* No prior history of chemotherapy and/or radiotherapy
* Able to read and understand either English or Mandarin

Exclusion Criteria:

* Physically or mentally unable to provide verbal/written consent
* Symptomatically ill (such as infection or an allergic reaction to chemotherapy)
* Presence of another condition for which fatigue is a prominent symptom (e.g. AIDS, fibromyalgia, or rheumatoid arthritis)
* Newly started on any medications that can cause general fatigue and body weakness (e.g. a beta-blocker or antidepressant, antihistamine, or antipsychotic medication)
* Presence of neurologic or immune-related medical condition or behavior known to influence the immune system (e.g. smoking or heavy drinking)

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The proposed study will be a multicenter, prospective, longitudinal, observational study conducted at the National Cancer Centre Singapore (NCCS) and KK Women's and Children's Hospital (KKH).
Sampling Method: Non-Probability Sample
Enrollment: 194 (Estimated)
Dates: Start 2014-10; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of cancer-related fatigue | One year post chemotherapy
  MFSI-SF will be used. This is a multidimensional questionnaire for measuring fatigue in cancer patients that has been validated in a group of breast cancer patients undergoing anticancer treatment. It consists of 30 items and has five subscales, each with six items: general fatigue, physical fatigue, emotional fatigue, mental fatigue, and vigor. The MFSI-SF measures different dimensions of fatigue, which can be combined to obtain an overall score. It has favorable psychometric properties with internal consistency reliability within the range of 0.87 to 0.96 and established convergent and divergent validity. As such, it is an appropriate tool for measuring fatigue.

SECONDARY OUTCOMES:
Incidence of cognitive impairment | One year post chemotherapy
  FACT-Cog will be used. The FACT-Cog was created to investigate the perceived impact of chemotherapy on cognitive functioning and associated impairments in quality of life. It is known in studies to assess broader aspects of cognitive complaints, thereby providing greater information about the types of cognitive complaints patients are experiencing. The qualitative data were examined using a thematic content analysis and the following domains were identified: Cognitive Problems (Cognitive), Impact on Functioning (IOF), and Impact on Quality of Life (QOL). Fifty items were written to assess these domains.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandre Chan, Singapore, Singapore